CLINICAL TRIAL: NCT07380412
Title: A Study to Evaluate the Effects of a Supplement on the Side Effects Associated With Stimulant Medications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Outliers, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20764
Record Dates: First submitted 2025-11-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Sleep Disturbance; Brain Fog
Keywords: ADHD; Anxiety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias; Mental Fatigue; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stasis Supplement (Experimental)
  Interventions: Dietary Supplement: Stasis Daytime and Nighttime
- Placebo Comparator (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Stasis Daytime and Nighttime — Daytime taken with stimulant medication and food. Nighttime taken 30 minutes before bedtime on an empty stomach.
  Arms: Stasis Supplement
Dietary Supplement: Placebo — Matched placebo product in taste and appearance.
  Arms: Placebo Comparator

SUMMARY:
This is a hybrid, two-arm, triple-blind, placebo-controlled, randomized clinical trial evaluating the efficacy of the Stasis supplement on reducing oxidative stress, cortisol levels, and side effects associated with stimulant medications used for ADHD over a three-month period in adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Currently prescribed stimulant medication for ADHD
* Experiencing: sleep difficulty, irritability, anxiety, brain fog
* Stable medication dose ≥3 months
* Healthy with no uncontrolled chronic conditions
* Stable on supplements ≥3 months if applicable
* US resident
* Willing to maintain current habits

Exclusion Criteria:

* Chronic conditions (e.g. cancer, mental illness)
* Use of psychiatric medications besides stimulants
* Pregnancy, breastfeeding, thyroid, liver, kidney conditions
* Recent smokers or heavy alcohol use
* Night shift workers
* Participation in other clinical trials
* Allergies to product ingredients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in oxidative stress and cortisol levels as measured by hs-CRP, 8-OHdG | Baseline and Month 3
  Measurement of oxidative stress and cortisol levels will be assessed using the following validated biomarkers:
  hs-CRP and serum cortisol from blood samples 8-hydroxy-2'-deoxyguanosine (8-OHdG) from urine samples
Change in cortisol levels | Baseline and Month 3
  Serum cortisol concentration measured via blood draw.

SECONDARY OUTCOMES:
Change in sleep quality | Baseline, Month 1, Month 2, and Month 3
  Sleep quality assessed via self-report questionnaire.
Change in irritability | Baseline, Month 1, Month 2, and Month 3
  Irritability assessed via self-report questionnaire.
Change in focus | Baseline, Month 1, Month 2, and Month 3
  Focus assessed via self-report questionnaire.
Change in sociability | Baseline, Month 1, Month 2, and Month 3
  Sociability assessed via self-report questionnaire.
Change in self-reported mood | Baseline, Month 1, Month 2, and Month 3
  Mood assessed via self-report questionnaire.
Change in self-reported stress | Baseline, Month 1, Month 2, and Month 3
  Stress levels assessed via self-report questionnaire.
Change in self-reported appetite | Baseline, Month 1, Month 2, and Month 3
  Appetite assessed via self-report questionnaire.
Change in blood levels of Vitamin C | Baseline and Month 3
  Serum levels of Vitamin C measured via blood test.
Change in blood levels of CoQ10 | Baseline and Month 3
  Serum levels of Coenzyme Q10 measured via blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States